CLINICAL TRIAL: NCT03064984
Title: Blood Based Eyedrops From Different Sources in the Treatment of Severe Keratopathy - A Randomized Clinical Trial
Brief Title: Blood Based Eyedrops From Different Sources in the Treatment of Severe Keratopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other); Regione Emilia-Romagna (Other); Centro Nazionale Sangue (Other Government)
Responsible Party: Principal Investigator, Emilio C Campos, Full Professor of Ophthalmology, Head Ophthalmology Unit, University of Bologna, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100/2016/O/Sper
Record Dates: First submitted 2017-02-15; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Keratopathy; Sjogren's Syndrome; GVHD - Graft-Versus-Host Disease
MeSH Terms: conditions — Sjogren's Syndrome; Graft vs Host Disease

STUDY DESIGN:
Intervention Model Description: This is a double-blind, interventional clinical study, randomized, multicenter. The treatments under study comprise topical products prepared from two different sources: umbilical cord blood collected at birth and adult subject donor peripheral blood. The products are prepared, standardized, controlled and sealed in anonymous frozen vials in the Transfusional Service, partner in the study.
  The study consists of two phases: Phase 1 is runned for one month treatment. The assignment of the treatment in Phase 1 is performed through a computer based randomization process, blind to the patient and the clinician, only known to the Transfusion Service personnel. The patient enter Phase 2 only in case of a corneal epithelial damage relapse taking place within two months after the end of Phase 1, and the treatment assigned belongs to the remaining arm. In this case also, the treatment is only known to the Transfusion Service personnel, trained to keep data aside.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The products under study are prepared, standardized, controlled and sealed in anonymous frozen vials in the Transfusional Service of the S.Orsola-Malpighi Hospital, our partner and collaborator in the study. The products have same physical and colour characteristics and cannot be visually recognized. Boxes containing the vials report a code of assignement only known by the Transfusion service personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBS eyedrops (Active Comparator): Eyedrops prepared from CBS (Cord Blood Serum), and administered 1 drop/each eye/8 times per day, for 30 days
  Interventions: Other: PBS eyedrops
- PBS eyedrops (Active Comparator): Eyedrops prepared from PBS (Peripheral Blood Serum) from adult donor subjects, administered 1 drop/each eye/8 times per day, for 30 days
  Interventions: Other: CBS eyedrops

INTERVENTIONS:
Other: CBS eyedrops — CBS eyedrops (prepared from umbilical cord blood serum) will be provided as frozen vials containing 0.8 ml of the product and will be administered at a regimen of 1 drop / 8 times day / each eye during the waking period, with the last administration to take before bedtime.
  Arms: PBS eyedrops
Other: PBS eyedrops — PBS eyedrops (prepared from adult peripheral blood serum) will be provided as frozen vials containing 0.8 ml of the product and will be administered at a regimen of 1 drop / 8 times day / each eye during the waking period, with the last administration to take before bedtime.
  Arms: CBS eyedrops

SUMMARY:
Topical preparations (eye drops) derived from the blood have become a relatively common treatment for more advanced forms of keratopathy. The purpose of this study is to evaluate the effect of two blood components from donors (serum cord blood and serum from adult subject donor peripheral blood) in the treatment of severe keratopathies.

DETAILED DESCRIPTION:
The rationale for the use of eye drops prepared from the blood as a source is mainly based on their content in growth factors (Growth factors, GF), which play an important role in regulation of many processes involved in normal healing of damaged corneal epithelium . The most used product so far is the eye drop prepared from serum (Autologous Serum, AS) or from platelet-rich plasma (Plasma Rich Platelet, PRP) of peripheral blood taken from the patients themselves. More recently, treatments were introduced by homologous sources that undoubtedly offer advantages as compared to autologous sources. In particular the homologous sources show:

* not invasiveness to the patient, who could in time not like the repeated withdrawals
* applicability even in patients with underlying systemic conditions. They may contain in their blood, among others, higher levels of pro-inflammatory factors, with the consequence of poor and inappropriate final product to be prepared and delivered to the eye

  * reliability, since the homologous products can be prepared, controlled, also validated under the microbiological profile and standardized advance, then kept frozen until the dispensation
  * conceptually unlimited availability of the product to be dispensed
  * versatility of therapeutic indications, based on different GF levels which are estimated in advance

The purpose of this study is to evaluate the effect of two products derived from two different blood sources (cord blood collected at birth from placenta umbilical veins and adult subject donor peripheral blood) in the treatment of severe keratopathies.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe dry eye , scored as level severity 3 according to the Dry Eye WorkShop grade (DEWS, Ocular Surf 2007)
* corneal epithelial damage, stained with fluorescein as vital dye, NEI (national Eye Institute) score> 6 (estimated with imageJ software) damage coverage> 25% of total corneal area
* good general health condition
* ability to adhere to treatment and to the procedures provided by the study

Exclusion Criteria:

* concurrent treatment with hypotensive drugs
* ocular surgery in the 12 months preceding enrollment .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Variation of corneal epithelium damage | 30 days
  The effect of the treatment(s) will be evaluated by measuring the area of damaged corneal epithelium (calculated as the mm2 of damaged epithelium) after treatment as compared to baseline, and defined as 1. complete healing : no detection of damaged area; 2. Partial healing : reduction of the damaged corneal area after treatment as compared to baseline ; 3. No improvement : same damaged corneal epithelial area in mm2 at baseline and after treatment; 4. Worsening : damaged corneal epithelial area in mm2 after treatment larger than at baseline

SECONDARY OUTCOMES:
Variation of subjective sensation of discomfort | 30 days
  The effect of the treatment(s) will be evaluated by measuring the subjective discomfort (expressed with the OSDI score) after treatment as compared to baseline and defined as 1. Disappearance of discomfort: OSDI score < 6/100; 2. Reduction of discomfort: reduction of the OSDI score after treatment as compared to baseline ; 3. No improvement : same values for OSDI score after treatment as detected in baseline; 4. Worsening : score for OSDI score after treatment higher than that detected at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emilio C Campos, MD, Principal Investigator — AOU Bologna, University of Bologna
Locations (3):
- Italy (3):
  - AOU Bologna, Ophthalmology Unit, Bologna, Bologna
  - Ospedale S.Maria Nuova - IRCCS - Ophthalmology Unit, Reggio Emilia, Reggio Emilia
  - Ospedale degli Infermi, Ophtalmology Unit, Rimini, Rimini

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Setten GB, Tervo T, Tervo K, Tarkkanen A. Epidermal growth factor (EGF) in ocular fluids: presence, origin and therapeutical considerations. Acta Ophthalmol Suppl (1985). 1992;(202):54-9. doi: 10.1111/j.1755-3768.1992.tb02169.x. No abstract available. PMID 1322012
- [Background] Marquez De Aracena Del Cid R, Montero De Espinosa Escoriaza I. Subconjunctival application of regenerative factor-rich plasma for the treatment of ocular alkali burns. Eur J Ophthalmol. 2009 Nov-Dec;19(6):909-15. doi: 10.1177/112067210901900603. PMID 19882589
- [Background] Ogawa Y, Okamoto S, Mori T, Yamada M, Mashima Y, Watanabe R, Kuwana M, Tsubota K, Ikeda Y, Oguchi Y. Autologous serum eye drops for the treatment of severe dry eye in patients with chronic graft-versus-host disease. Bone Marrow Transplant. 2003 Apr;31(7):579-83. doi: 10.1038/sj.bmt.1703862. PMID 12692625
- [Background] Tsubota K, Goto E, Fujita H, Ono M, Inoue H, Saito I, Shimmura S. Treatment of dry eye by autologous serum application in Sjogren's syndrome. Br J Ophthalmol. 1999 Apr;83(4):390-5. doi: 10.1136/bjo.83.4.390. PMID 10434857
- [Background] Lopez-Plandolit S, Morales MC, Freire V, Etxebarria J, Duran JA. Plasma rich in growth factors as a therapeutic agent for persistent corneal epithelial defects. Cornea. 2010 Aug;29(8):843-8. doi: 10.1097/ICO.0b013e3181a81820. PMID 20508516
- [Background] Yoon KC, Im SK, Park YG, Jung YD, Yang SY, Choi J. Application of umbilical cord serum eyedrops for the treatment of dry eye syndrome. Cornea. 2006 Apr;25(3):268-72. doi: 10.1097/01.ico.0000183484.85636.b6. PMID 16633024
- [Background] Yoon KC, You IC, Im SK, Jeong TS, Park YG, Choi J. Application of umbilical cord serum eyedrops for the treatment of neurotrophic keratitis. Ophthalmology. 2007 Sep;114(9):1637-42. doi: 10.1016/j.ophtha.2006.12.014. Epub 2007 Mar 26. PMID 17382396
- [Background] Yoon KC, Choi W, You IC, Choi J. Application of umbilical cord serum eyedrops for recurrent corneal erosions. Cornea. 2011 Jul;30(7):744-8. doi: 10.1097/ICO.0b013e31820d850f. PMID 21436685
- [Background] Sharma N, Goel M, Velpandian T, Titiyal JS, Tandon R, Vajpayee RB. Evaluation of umbilical cord serum therapy in acute ocular chemical burns. Invest Ophthalmol Vis Sci. 2011 Feb 25;52(2):1087-92. doi: 10.1167/iovs.09-4170. PMID 20538982
- [Background] Versura P, Profazio V, Buzzi M, Stancari A, Arpinati M, Malavolta N, Campos EC. Efficacy of standardized and quality-controlled cord blood serum eye drop therapy in the healing of severe corneal epithelial damage in dry eye. Cornea. 2013 Apr;32(4):412-8. doi: 10.1097/ICO.0b013e3182580762. PMID 22955120
- [Background] Versura P, Buzzi M, Giannaccare G, Grillini M, Terzi A, Pagliaro P, Campos EC. Cord blood serum-based eye drops: the impact of donor haematological and obstetric factors on the variability of epidermal growth factor levels. Blood Transfus. 2014 Jan;12 Suppl 1(Suppl 1):s44-50. doi: 10.2450/2013.0115-13. Epub 2013 Oct 3. PMID 24120597
- [Background] Versura P, Buzzi M, Giannaccare G, Terzi A, Fresina M, Velati C, Campos EC. Targeting growth factor supply in keratopathy treatment: comparison between maternal peripheral blood and cord blood as sources for the preparation of topical eye drops. Blood Transfus. 2016 Mar;14(2):145-51. doi: 10.2450/2015.0020-15. Epub 2015 Jul 9. PMID 26192781
- [Background] van der Meer PF, Seghatchian J, de Korte D. Autologous and allogeneic serum eye drops. The Dutch perspective. Transfus Apher Sci. 2015 Aug;53(1):99-100. doi: 10.1016/j.transci.2015.05.017. Epub 2015 Jun 9. PMID 26138910
- [Background] Espinosa A, Hjorth-Hansen H, Aasly K, Teigum I, Sivertsen G, Seghatchian J. Implementation of a standardised method for the production of allogeneic serum eye drops from regular blood donors in a Norwegian University Hospital: Some methodological aspects and clinical considerations. Transfus Apher Sci. 2015 Aug;53(1):88-91. doi: 10.1016/j.transci.2015.05.014. Epub 2015 May 19. PMID 26027793
- [Background] Harritshoj LH, Nielsen C, Ullum H, Hansen MB, Julian HO. Ready-made allogeneic ABO-specific serum eye drops: production from regular male blood donors, clinical routine, safety and efficacy. Acta Ophthalmol. 2014 Dec;92(8):783-6. doi: 10.1111/aos.12386. Epub 2014 Mar 16. PMID 24629028
- [Background] Adelman SF, Howett MK, Rapp F. Protease inhibitors suppress fibrinolytic activity of herpesvirus-transformed cells. J Gen Virol. 1982 May;60(Pt 1):15-24. doi: 10.1099/0022-1317-60-1-15. PMID 6178796
- [Derived] Campos E, Versura P, Buzzi M, Fontana L, Giannaccare G, Pellegrini M, Lanconelli N, Brancaleoni A, Moscardelli F, Sebastiani S, Vaselli C, Randi V. Blood derived treatment from two allogeneic sources for severe dry eye associated to keratopathy: a multicentre randomised cross over clinical trial. Br J Ophthalmol. 2020 Aug;104(8):1142-1147. doi: 10.1136/bjophthalmol-2019-314859. Epub 2019 Nov 19. PMID 31744796